CLINICAL TRIAL: NCT03429946
Title: Hypoglycemia and Autonomic Nervous System Function
Brief Title: Hypoglycemia and Autonomic Nervous System Function-B
Acronym: HypoANS-B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Gail Kurr Adler, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2004P001233-B; R01HL109634 (NIH); K24HL103845 (NIH); UL1TR001102 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hypoglycemia; Healthy
MeSH Terms: conditions — Hypoglycemia | interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: Participants complete all 3 arms of the study in random order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigator performing the clamp studies is only aware of the type of clamp - euglycemic versus hypoglycemic - but not aware of placebo versus spironolactone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Hypoglycemia and Spironolactone (Active Comparator): Participants undergo two 120-minute hypoglycemic hyperinsulinemic clamp procedures (50 mg/dL) - an AM clamp from about 9 am to 11 am and a PM clamp from 1 pm to 3 pm on Day 2 of a 3-Day study visit. Participants receive two doses of 100 mg of spironolactone - one dose 12 hours and one dose 3 hours before the first clamp starts. Modified Oxford Procedure is performed in duplicate at six time points - on Day 1, before the AM hyperinsulinemic clamp, during the AM hyperinsulinemic clamp, before the PM hyperinsulinemic clamp, during the PM hyperinsulinemic clamp, and on Day 3. The Modified Oxford procedure is performed to calculate baroreflex sensitivity.
  Interventions: Drug: Spironolactone; Other: Hypoglycemic Hyperinsulinemic Clamp
- Hypoglycemia and Placebo (Active Comparator): Participants undergo two 120-minute hypoglycemic hyperinsulinemic clamp procedures (50 mg/dL) - an AM clamp from about 9 am to 11 am and a PM clamp from 1 pm to 3 pm on Day 2 of a 3-Day study visit. Participants receive two doses of placebo - one dose 12 hours and one dose 3 hours before the first clamp starts. Modified Oxford Procedure is performed in duplicate at six time points - on Day 1, before the AM hyperinsulinemic clamp, during the AM hyperinsulinemic clamp, before the PM hyperinsulinemic clamp, during the PM hyperinsulinemic clamp, and on Day 3. The Modified Oxford procedure is performed to calculate baroreflex sensitivity.
  Interventions: Drug: Placebo; Other: Hypoglycemic Hyperinsulinemic Clamp
- Euglycemia and Placebo (Placebo Comparator): Participants undergo two 120-minute euglycemic hyperinsulinemic clamp procedures (90 mg/dL) - an AM clamp from about 9 am to 11 am and a PM clamp from 1 pm to 3 pm on Day 2 of a 3-Day study visit. Participants receive two doses of placebo - one dose 12 hours and one dose 3 hours before the first clamp starts. Modified Oxford Procedure is performed in duplicate at six time points - on Day 1, before the AM hyperinsulinemic clamp, during the AM hyperinsulinemic clamp, before the PM hyperinsulinemic clamp, during the PM hyperinsulinemic clamp, and on Day 3. The Modified Oxford procedure is performed to calculate baroreflex sensitivity.
  Interventions: Drug: Placebo; Other: Euglycemic Hyperinsulinemic Clamp

INTERVENTIONS:
Drug: Spironolactone — Participants will receive spironolactone 12 hours and 3 hours before the initiation of the hyperinsulinemic clamp treatment.
  Arms: Hypoglycemia and Spironolactone
Drug: Placebo — Participants will receive placebo 12 hours and 3 hours before the initiation of the hyperinsulinemic clamp treatment.
  Arms: Euglycemia and Placebo; Hypoglycemia and Placebo
Other: Hypoglycemic Hyperinsulinemic Clamp — Participants undergo two 120-minute hypoglycemic (50 mg/dL) hyperinsulinemic clamps - an AM clamp from about 9 am to 11 am and a PM clamp from 1 pm to 3 pm on Day 2 of a 3-Day study visit. Modified Oxford Procedure is performed in duplicate at six time points - on Day 1, before the AM hyperinsulinemic clamp, during the AM hyperinsulinemic clamp, before the PM hyperinsulinemic clamp, during the PM hyperinsulinemic clamp, and on Day 3. The Modified Oxford procedure is performed to calculate baroreflex sensitivity.
  Other Names: Hypoglycemic Hyperinsulinemic Clamp Procedure
  Arms: Hypoglycemia and Placebo; Hypoglycemia and Spironolactone
Other: Euglycemic Hyperinsulinemic Clamp — Participants undergo two 120-minute euglycemic (90 mg/dL) hyperinsulinemic clamps - an AM clamp from about 9 am to 11 am and a PM clamp from 1 pm to 3 pm on Day 2 of a 3-Day study visit.Modified Oxford Procedure is performed in duplicate at six time points - on Day 1, before the AM hyperinsulinemic clamp, during the AM hyperinsulinemic clamp, before the PM hyperinsulinemic clamp, during the PM hyperinsulinemic clamp, and on Day 3. The Modified Oxford procedure is performed to calculate baroreflex sensitivity.
  Other Names: Euglycemic Hyperinsulinemic Clamp Procedure
  Arms: Euglycemia and Placebo

SUMMARY:
This study tests the hypothesis that, compared to prior normal blood sugar, prior low blood sugar impairs cardiovascular autonomic function. The proposed studies will also test the hypothesis that the effects of prior low blood sugar on cardiovascular autonomic function are blocked by administration of a mineralocorticoid receptor antagonist.

DETAILED DESCRIPTION:
This study involves three interventions, which are performed in random order. Each intervention involves a 3-day inpatient visit. There is a space of 1-3 months between interventions. The three interventions are: 1) placebo with a hyperinsulinemic euglycemic clamp, 2) spironolactone with a hyperinsulinemic hypoglycemic clamp, or 3) placebo with a hyperinsulinemic hypoglycemic clamp. Each 3-day inpatient visit includes the following. On Day 1, autonomic testing is performed. Autonomic testing includes assessment of Baroreflex Sensitivity (BRS). BRS is assessed using the Modified Oxford procedure, which involves sequential administration of nitroprusside and phenylephrine while measuring heart rate and beat to beat blood pressure with a finapress and assessing Muscle Sympathetic Nerve Activity (MSNA). MSNA is measured using microelectrodes placed near the peroneal nerve. On Day 2, hyperinsulinemic clamps are performed with pre-treatment with either placebo or spironolactone. Modified Oxford Procedures are performed prior to and during each clamp on Day 2. On Day 3, the autonomic testing performed on Day 1 is repeated..

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Males and females age 18 to 55 years

Exclusion Criteria:

* Pregnancy
* Lactation
* Clinically evident coronary artery, cerebrovascular, or peripheral vascular disease, or presence of systemic illness that might affect autonomic function. Such illnesses include diabetes mellitus, congestive heart failure, hypertension, renal, pulmonary, hepatic disease, anemia, malignancies, untreated thyroid disease, and alcoholism.
* Current major depressive illness
* In all subjects, any individuals on oral, injected, inhaled or topical corticosteroids within the last year or oral contraceptives within the past 3 months will be excluded.
* Use of medications other than thyroxine
* Known hypersensitivity to nitroglycerin, nitroprusside and/or phenylephrine.
* Blood pressure > 140/90 mmHg
* Creatinine > 1.5 mg/dL
* Serum potassium >5.2 mmol/L
* Estimated GFR < 50 mL/min
* Use of Viagra, Cialis, and similar drugs within 72 hours of admission.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Baroreflex Sensitivity assessed on Day 3 | Baroreflex sensitivity is assessed on the 3rd day of each treatment (i.e. about 16 hours after completion of the hyperinsulinemic clamp)
  Comparison of Day 3 baroreflex sensitivity (milliseconds/mm Hg) assessed during Hypoglycemic hyperinsulinemic clamp + Placebo treatment as compared to Hypoglycemic hyperinsulinemic clamp + Spironolactone treatment.

SECONDARY OUTCOMES:
Muscle sympathetic nerve activity assessed on Day 3 | Muscle sympathetic nerve activity is assessed on the 3rd day of each treatment (i.e. about 16 hours after completion of the hyperinsulinemic clamp)
  Comparison of Day 3 muscle sympathetic nerve activity (bursts/min) assessed during hypoglycemic hyperinsulinemic clamp + placebo treatment as compared to hypoglycemic hyperinsulinemic clamp + spironolactone treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Adler, MD/PhD, Principal Investigator — Brigham and Women's Hospital; Roy Freeman, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The data collected will comply with the NIH requirements for timely release and data sharing. Data will be shared in the form of publications and presentations in scientific forums. As the NIH has noted, the investigators reserve the right to keep the data restricted in order to perform the initial analyses for this grant proposal and will continue to use the data for further, but not prolonged, exclusive use. Of note, the sharing of this data will be limited by at least the following issues, some unique to this proposal and some not unique. Some of the data obtained in this study is defined to be sensitive in nature, which may restrict its ability to be shared. Data may only be shared with the approval of our IRB and is limited by HIPPA and any other regulations that may be promulgated during the course of this proposal.
Time Frame: Data will be shared after completion of study and initial publications which we anticipate to be within 18 months of the final participant completing the study protocol.
Access Criteria: Access to data must be approved by the IRB at our institution.